CLINICAL TRIAL: NCT02002715
Title: Randomised, Open-label, Parallel-group Study of Therapeutic Effect of Different Treatment Course With Inhaled Corticosteroids in Eosinophilic Bronchitis Patients
Brief Title: Therapeutic Effect of Different Treatment Course With Inhaled Corticosteroids in Eosinophilic Bronchitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cough001
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Eosinophilic Bronchitis
Keywords: eosinophilic bronchitis; inhaled corticosteroids; therapeutic effect
MeSH Terms: interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inhaled budesonide for 4 weeks (Active Comparator): inhaled Budesonide 100µg , 2puff Q12h for 4 weeks
  Interventions: Drug: Inhaled budesonide
- Inhaled budesonide for 8 weeks (Active Comparator): inhaled Budesonide 100µg , 2puff Q12h for 8 weeks
  Interventions: Drug: Inhaled budesonide
- Inhaled budesonide for 16 weeks (Active Comparator): inhaled Budesonide 100µg , 2puff Q12h for 16 weeks
  Interventions: Drug: Inhaled budesonide

INTERVENTIONS:
Drug: Inhaled budesonide — inhaled Budesonide 2puff Q12h,total 400µg/day for 4 weeks inhaled Budesonide 2puff Q12h,total 400µg/day for 8 weeks inhaled Budesonide 2puff Q12h,total 400µg/day for 16 weeks
  Other Names: Budesonide Powder for Inhalation

SUMMARY:
This study aims to observe the therapeutic effect of different treatment course with inhaled corticosteroids in eosinophilic bronchitis patients.

The investigators hypothesize:

1. Cough score will be improved after treatment with longer treatment course with inhaled corticosteroids in EB patients.
2. The sputum eosinophil percentage will be decreased and recovered to normal level (Eos%<2.5%) with longer treatment course with inhaled corticosteroids in EB patients.
3. The rate of recurrence after treatment will be decrease with longer treatment course with inhaled corticosteroids in EB patients

DETAILED DESCRIPTION:
Study groups:

Patients diagnosed with EB will be randomised into three groups as follows:

Group 1(4-week treatment group):The patients with eosinophilic bronchitis received Pulmicourt Turbuhaler (Budesonide 100µg) 2puff Q12h for 4 weeks.

Group 2(8-week treatment group):The patients with eosinophilic bronchitis received Pulmicourt Turbuhaler (Budesonide 100µg) 2puff Q12h for 8 weeks.

Group 3(16-week treatment group):The patients with eosinophilic bronchitis received Pulmicourt Turbuhaler (Budesonide 100µg) 2puff Q12h for 16 weeks.

The study will be divided into following phases:

1. First Visit (Visit 1, day -3):

   A full medical history and physical examination to be undertaken to determine whether patients meet the inclusion/exclusion criteria.

   After the informed consent has been signed, the following samples are obtained from all patients: blood samples for routine clinical laboratory tests (haematology, biochemistry and chest x-ray). A urine pregnancy test will be performed in women of childbearing potential.

   Bronchial provocation test by methacholine inhalation are performed to determined whether it presences of bronchial non-specific hyper-responsiveness. Hypertonic saline induced sputum samples for cell differential is taken to determine whether it esixt eosinophilic airway inflammation.
2. Second Visit (Visit 2, Week 0):

   A physical examination was to be performed. All laboratory tests results are obtained to determine whether patients meet the inclusion/exclusion criteria. Enrolled patients are randomly divided into three groups with inhaled budesonide 200 µg twice daily via a turbohaler for 4 weeks, 8 weeks and 16 weeks respectively and given the Diary Card.
3. During Treatment (Week 0 to Week 4/8/16,every 4 weeks):

   Patients were to take study medication for 4 weeks in 4-week group,8 weeks in 8-week group,16 weeks in 16-week group. All patient are followed-up every 4 weeks and completed Diary Card for 7 days in the last week of treatment.
4. Third Visit (Visit 3, Week 4/8/16):

   A physical examination were to be performed. The Diary Card were collected and reviewed. Adverse events, secondary complications, concurrent medication will be recorded.Hypertonic saline induced sputum samples for cell differential is taken from enrolled patients.Blood samples for routine clinical laboratory tests (haematology and biochemistry) were obtained
5. Follow-up visits were conducted after 1 year and whenever recurrence of cough :Cough symptom score,visual analogue scale (VAS), spiromery and induced sputum for cell differential is taken from enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a history of cough as sole or main symptom lasting more than 3 weeks.
2. Patients whose chest x-ray outcome was normal or without any active focus.
3. Patients who were diagnosed with the result of sputum eosinophil percentage (Eos%) over 2.5%, and the negative result in bronchial provocation test by methacholine inhalation challenge.
4. Patients who was aged from 18 years old (≥ 18 years old ) to 75 years old (≤ 75 years old).

Exclusion Criteria:

1. Patients who is a smoker or ex-smoker and has smoked within the previous year or has a cumulative smoking history >10 pack-years or equivalence.
2. Patients with concomitance of GERC (gastroesophageal reflux-related chronic cough), chronic bronchitis , bronchiectasis, bronchial tuberculosis, ACEI induced cough, bronchogenic carcinoma, psychologic cough, pulmonary fibrosis, bronchus foreign body, microlithiasis, tracheobroncheopathia osteochondroplastica, mediastinal tumor, left ventricular dysfunction.
3. Female subjects who are pregnant, breast-feeding or risk of becoming pregnant during the study.
4. Subjects who are known or suspected to be hypersensitive to any component of the study medication or relief medications.
5. Subjects who have received any therapy in the previous 4 weeks, e.g.corticosteroids ,antihistamines, leukotriene receptor antagonist in previous 4 weeks
6. Subjects who are diagnosed with past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease. e.g.nasal-sinus infection, lower respiratory tract infection, chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis or bronchopulmonary dysplasia.
7. Subjects who demonstrate significant abnormality on biochemistry, hematology, ECG.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the relapse rate of eosinophilic bronchitis in one year. | 1 year

SECONDARY OUTCOMES:
change in percentage of eosinophil in induced sputum from baseline to post-treatment | week 0,week 4,week 8,week 16
change in Cough visual analogue scale (VAS) and Cough Symptom Score (CSS) from baseline to post-treatment | week 0,week 4,week 8,week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhan W, Tang J, Chen X, Yi F, Han L, Liu B, Luo W, Chen Q, Lai K. Duration of treatment with inhaled corticosteroids in nonasthmatic eosinophilic bronchitis: a randomized open label trial. Ther Adv Respir Dis. 2019 Jan-Dec;13:1753466619891520. doi: 10.1177/1753466619891520. PMID 31847717